CLINICAL TRIAL: NCT04792112
Title: Improving Clinical Practice Guidelines for Antenatal Corticosteroids: Incorporating a Decision Support Tool to Tackle the Uncertain Balance of Harms and Benefits
Brief Title: Navigating the Grey Zone for Antenatal Corticosteroids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jessica Liauw, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H20-03071
Record Dates: First submitted 2021-02-25; First posted 2021-03-10 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Decision Making, Shared; Pregnancy; Preterm Birth
Keywords: Antenatal corticosteroid
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Controlled before and after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guideline + decision support tool (Experimental): A decision support tool summarizing harms and benefits of late preterm antenatal corticosteroids will be integrated into the clinical practice guideline available to clinicians in the hospitals in the experimental arm.
  Interventions: Behavioral: Decision support tool
- Guideline only (No Intervention): Clinicians in the hospitals in the 'no-intervention' arm will have access to the standard guideline only (without the integrated decision support tool).

INTERVENTIONS:
Behavioral: Decision support tool — Decision support tool for late preterm antenatal corticosteroids
  Arms: Guideline + decision support tool

SUMMARY:
The purpose of this study is to find out if including a decision support tool in clinical practice guidelines will improve how doctors discuss the option of antenatal corticosteroid treatment with patients who might deliver at 34 to 36 weeks of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 year or older.
* Delivered a live neonate at 34+0 to 36+6 weeks of gestation.
* Speaks English.
* Agrees to participate in the questionnaire during their first week post-partum.
* Delivered at one of the six participating obstetrical hospitals.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
The change in frequency of clinical counselling about late preterm antenatal corticosteroids. | up to 8 months following implementation of the intervention.
  The difference in the proportion of patients who delivered a neonate at 34+0 to 36+6 weeks' gestation who report having had a discussion about antenatal corticosteroids with their care provider pre-intervention versus post-intervention.

SECONDARY OUTCOMES:
The change in quality of clinical counselling about late preterm antenatal corticosteroids as assessed by the COMRADE scale. | up to 8 months following implementation of the intervention.
  The difference in the average median score on the Combined Outcome Measure for Risk Communication and Treatment Decision Making Effectiveness (COMRADE) scale, among those that report having had a discussion about late preterm antenatal corticosteroids with their health care provider. We will use an adapted scale including 19 items, each of which are scored on a 5-point Likert scale. A higher score indicates better risk communication and treatment decision making effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Liauw, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Surrey Memorial Hospital, Surrey, British Columbia
  - BC Women's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No